CLINICAL TRIAL: NCT04684199
Title: The Therapeutic Effect of Melatonin in Pediatric Patients With Functional Dyspepsia
Brief Title: Melatonin in Pediatric FD Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14010042
Record Dates: First submitted 2014-07-23; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Dyspepsia
Keywords: Functional Dyspepsia; Melatonin; Pain; Actigraphy and Pain
MeSH Terms: conditions — Dyspepsia; Pain | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator): Melatonin
  All participants will receive a 5 mg. dose of melatonin before bed for a period of two weeks during study period.
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): Placebo
  All participants will receive a placebo comparative in substance, color, and flavor, before bed for two weeks during the study.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Comparison between melatonin and placebo (2 weeks each) with active and placebo crossover during the study period of 34-36 days.
  Other Names: Melatonin 5 mg.
  Arms: Melatonin
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
There are two specific aims in this study.

Specific Aim 1: Determine if melatonin results in a higher grade of clinical response than does placebo in children with functional dyspepsia (FD).

Hypothesis: treatment of FD with melatonin will result in a higher grade of clinical response than will treatment with a placebo.

Specific Aim 2: Evaluate the relationship between changes in sleep and improvement in pain in pediatric patients with functional dyspepsia receiving melatonin.

Hypothesis: There will be no association between improvement in pain and improvement in sleep in children with functional dyspepsia receiving melatonin.

DETAILED DESCRIPTION:
Recurrent abdominal pain is present in a significant proportion of the pediatric population at large. Often times, no clear organic cause for pain will be found, and these children are diagnosed with functional abdominal pain. Of the children with functional abdominal pain, many are classified as having functional dyspepsia (FD). Functional dyspepsia is defined as persistent or recurrent pain or discomfort centered in the upper abdomen (above the umbilicus) that is unrelated to a change in stool frequency or form and not exclusively relieved by defecation. There have been only a few placebo controlled trials of medications in children with abdominal pain and none in children specifically with functional dyspepsia and uninvestigated mucosal inflammation.

There is increasing evidence suggesting that melatonin plays a role in pain modulation. Melatonin is produced by the pineal gland and is recognized for its regulation of sleep and circadian functions. Less widely recognized is melatonin's production in other parts of the body; such as in the digestive system and in immune cells including mast cells. The total amount of melatonin in the digestive system exceeds that of the pineal gland and blood. Within the digestive tract, melatonin is produced in the enterochromaffin cells. It exerts both excitatory and inhibitory effects on the enteric nervous system as well as possessing anti-inflammatory and immunomodulatory properties. In a rat model of reflux esophagitis, melatonin demonstrated multiple effects on the esophageal mucosa. These included decreased lipid peroxidation (oxidative degradation of lipids in cell membranes which leads to cell damage), replenished superoxide dismutase and glutathione (improved defense of the mucosa), and decreased expression of T helper 1 cytokines (pro-inflammatory cytokines) while not altering anti inflammatory cytokines. These effects may account for the reduction in pain in adults with irritable bowel syndrome (IBS) and dyspepsia during a trial of melatonin therapy. In a study of adults with IBS in association with sleep disturbances, patients were given melatonin 3mg or placebo at bedtime for two weeks. Compared with the placebo group, the group who received melatonin had significantly lower mean abdominal pain scores while sleep parameters were not influenced. In a study of adults with functional dyspepsia, twelve weeks of melatonin (5 mg taken at bedtime) resulted in 56.6% of patients having complete resolution of symptoms and 30% having partial improvement, while only 6.7% of the patients who received placebo experienced any improvement in symptoms. Melatonin has not been previously studied in children with abdominal pain. Evaluation of its effects is warranted as melatonin would be a very safe and inexpensive alternative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the GI clinic with a diagnosis of functional dyspepsia as defined by Rome III criteria.
* Persistent pain despite acid suppression at therapeutic doses for at least 4 weeks
* Patients ages 8-17 years, inclusive.

Exclusion Criteria:

* Patients currently using melatonin.
* Patients who have previously had endoscopy.
* Initiation of a treatment plan that includes one or more of the following medications in the last 4 weeks

  * Opiates
  * Tramadol
  * Gabapentin
  * Benzodiazepines

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Grade of clinical response to Melatonin in children with functional dyspepsia | 35 days
  The overall positive response rate (grade 3-5) will be compared between melatonin and placebo by the McNemar test.

SECONDARY OUTCOMES:
Change in sleep in pediatric patients with functional dyspepsia receiving melatonin | 35 days
  The mean sleep latency and mean sleep duration from sleep diary and actigraphy data will be compared between baseline and therapy for melatonin and placebo, respectively, using the paired Student's t test.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sturgeon, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] APLEY J, NAISH N. Recurrent abdominal pains: a field survey of 1,000 school children. Arch Dis Child. 1958 Apr;33(168):165-70. doi: 10.1136/adc.33.168.165. No abstract available. PMID 13534750
- [Background] Rasquin-Weber A, Hyman PE, Cucchiara S, Fleisher DR, Hyams JS, Milla PJ, Staiano A. Childhood functional gastrointestinal disorders. Gut. 1999 Sep;45 Suppl 2(Suppl 2):II60-8. doi: 10.1136/gut.45.2008.ii60. PMID 10457047
- [Background] Shaffer SE, Sellman SB, Repucci AH, Hupertz VF, Czinn SJ, Boyle JT. Dyspepsia: Redefining chronic abdominal pain in children. Gastroenterology. 1992; 102:163A
- [Background] Ambriz-Tututi M, Rocha-Gonzalez HI, Cruz SL, Granados-Soto V. Melatonin: a hormone that modulates pain. Life Sci. 2009 Apr 10;84(15-16):489-98. doi: 10.1016/j.lfs.2009.01.024. Epub 2009 Feb 15. PMID 19223003
- [Background] Maldonado MD, Mora-Santos M, Naji L, Carrascosa-Salmoral MP, Naranjo MC, Calvo JR. Evidence of melatonin synthesis and release by mast cells. Possible modulatory role on inflammation. Pharmacol Res. 2010 Sep;62(3):282-7. doi: 10.1016/j.phrs.2009.11.014. Epub 2009 Dec 4. PMID 19963060
- [Background] Klupinska G, Poplawski T, Drzewoski J, Harasiuk A, Reiter RJ, Blasiak J, Chojnacki J. Therapeutic effect of melatonin in patients with functional dyspepsia. J Clin Gastroenterol. 2007 Mar;41(3):270-4. doi: 10.1097/MCG.0b013e318031457a. PMID 17426465
- [Background] Song GH, Leng PH, Gwee KA, Moochhala SM, Ho KY. Melatonin improves abdominal pain in irritable bowel syndrome patients who have sleep disturbances: a randomised, double blind, placebo controlled study. Gut. 2005 Oct;54(10):1402-7. doi: 10.1136/gut.2004.062034. Epub 2005 May 24. PMID 15914575
- [Background] Lahiri S, Singh P, Singh S, Rasheed N, Palit G, Pant KK. Melatonin protects against experimental reflux esophagitis. J Pineal Res. 2009 Mar;46(2):207-13. doi: 10.1111/j.1600-079X.2008.00650.x. Epub 2008 Nov 28. PMID 19067786
- [Background] Buck M. The Use of Melatonin in Children With Sleep Disturbances. Pediatr Pharm. 2003;9(11)
- [Background] Kobayashi I, Hall B, Palmieri P. Acigraphy improves measurements of sleep functioning. Traumatic Stress Points. 2008 Mar Vol 22, Issue 2
- [Background] Meltzer LJ, Montgomery-Downs HE, Insana SP, Walsh CM. Use of actigraphy for assessment in pediatric sleep research. Sleep Med Rev. 2012 Oct;16(5):463-75. doi: 10.1016/j.smrv.2011.10.002. Epub 2012 Mar 15. PMID 22424706
- [Background] Cellini N, Buman MP, McDevitt EA, Ricker AA, Mednick SC. Direct comparison of two actigraphy devices with polysomnographically recorded naps in healthy young adults. Chronobiol Int. 2013 Jun;30(5):691-8. doi: 10.3109/07420528.2013.782312. Epub 2013 May 30. PMID 23721120
- [Background] Sadeh A, Sharkey KM, Carskadon MA. Activity-based sleep-wake identification: an empirical test of methodological issues. Sleep. 1994 Apr;17(3):201-7. doi: 10.1093/sleep/17.3.201. PMID 7939118
- [Background] Weiss MD, Wasdell MB, Bomben MM, Rea KJ, Freeman RD. Sleep hygiene and melatonin treatment for children and adolescents with ADHD and initial insomnia. J Am Acad Child Adolesc Psychiatry. 2006 May;45(5):512-519. PMID 16670647